CLINICAL TRIAL: NCT00317564
Title: Betaseron Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Syneos Health (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 308740
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Birth Defects; Pregnancy Complications; Multiple Sclerosis
Keywords: Birth Defects; High Risk Pregnancy; Multiple Sclerosis
MeSH Terms: conditions — Congenital Abnormalities; Pregnancy Complications; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective, observational, registration and follow-up study of women exposed to Betaseron® at the time of conception (i.e., any time from the first day of the last menstrual period) and/or during pregnancy. The Betaseron® Pregnancy Registry is designed to determine whether there is an increased risk or a pattern of birth defects in the offspring of women exposed to Betaseron® at conception and during pregnancy compared to rates from women in the general US population. Secondarily, the Registry will examine rates of spontaneous abortions and other negative pregnancy outcomes in this population. This study will be conducted in the United States (US). The Betaseron® Pregnancy Registry is sponsored by Bayer HealthCare Pharmaceuticals and is managed by the Post Approval & Strategic Services group at INC Research, LLC. The scientific conduct and analysis of the Registry will be overseen by an Independent Data Safety Monitoring Board (IDSMB) consisting of external specialists in teratology, epidemiology, maternal and fetal medicine, and neurology (external member details available upon request).

DETAILED DESCRIPTION:
Because informed consent is required, the Registration process must be initiated by the patient. An HCP who contacts the Registry may request an authorization for release of medical information packet or have the eligible patient contact the Registry directly. Once an eligible subject provides consent and permission to obtain information from her HCP, the Registry will contact the obstetric HCP and obtain information on demographics, history of previous pregnancies, maternal risk factors, pregnancy outcome, and neonatal health. Data will be collected from the maternal HCP at enrollment, during the second trimester (around week 20), and at outcome. Data on live born infants will be collected from the pediatrician at 4 months of age. If a birth defect is reported, targeted follow-up may be conducted.

NOTE: This study has previously been posted by Berlex, Inc. which has since been renamed to Bayer HealthCare Pharmaceuticals, Inc. Bayer HealthCare Pharmaceuticals, Inc. is the sponsor of this pregnancy registry.

ELIGIBILITY:
Inclusion Criteria:

The subjects must meet the following criteria for registration:

* Enroll prospectively (patient is still pregnant and no structural defects have been noted on a prenatal test)
* Diagnosed with MS prior to or during the current pregnancy
* Exposed to Betaseron® on or after the first day of the patient's last menstrual period
* Provide verbal consent to participate in the Registry
* Verbally provide contact information for herself, her HCP, and the infant's HCP (as applicable)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: US only
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2006-04; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Albano, PhD, MS, Principal Investigator — Syneos Health; Vicki Poon, MPH, Study Director — Bayer; Mark Rametta, D.O., FACOI, FACP, Study Director — Bayer; Karen Maloney Marini, Study Director — Bayer
Locations (1):
- INC Research, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Coyle PK, Sinclair SM, Scheuerle AE, Thorp JM Jr, Albano JD, Rametta MJ. Final results from the Betaseron (interferon beta-1b) Pregnancy Registry: a prospective observational study of birth defects and pregnancy-related adverse events. BMJ Open. 2014 May 12;4(5):e004536. doi: 10.1136/bmjopen-2013-004536. PMID 24821713